CLINICAL TRIAL: NCT02927561
Title: Automated Diagnostic Test for Diabetic Retinopathy in Brazilian Mass Screening
Status: Completed | Type: Observational
Sponsor: Retina Clinic, Sao Paulo, Brazil (Other)
Responsible Party: Sponsor
Other Study IDs: Retina C
Record Dates: First submitted 2016-09-30; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Diabetic Retinopathy screening — Diabetic Retinopathy screening

SUMMARY:
In Brazil 10% of the adult population has diabetes. Of these, 39.0% are undiagnosed, at risk for developing complications such as diabetic retinopathy (DR). Due to the increasing prevalence of diabetes and high percentage of patients with uncontrolled disease, cost-effective tools are needed with focused attention on diabetes prevention and management in the current health system. The automatic retinopathy detection can enlarge the screening, reducing the workload and costs compared to manual image graders.

DETAILED DESCRIPTION:
In the South and Central America Region, an estimated 9.4% of the adult population (20-79 years) has diabetes in 2015, and Brazil is the first country in number of people with diabetes. Of these, 39.0% are undiagnosed, at risk for developing complications such as diabetic retinopathy (DR)(1).

The rising number of people with diabetes in the world has become a real challenge for the public health system to provide care for patients with DR and for people with diabetes at risk for this complication(2). A large proportion of patients with diabetes was inadequately controlled in Brazil, which may contribute to increased rates of diabetic complications (3).

The detection of any degree of DR may result in improved medical monitoring and optimization of risk factors, delaying the progression of the disease(4). In Brazil, the great demand in the public service causes delay in early diagnosis, worsening health status of patients with diabetic retinopathy and increasing the cost of their treatment.

Due to the increasing prevalence of diabetes and high percentage of patients with uncontrolled disease, cost-effective tools are needed with focused attention on diabetes prevention and management in the current health system.

Several studies have shown that systematic screening for DR is an effective way of prevention (5). Furthermore, the automatic retinopathy detection can enlarge the screening, reducing the workload and costs compared to manual image graders(6). There are no reports on automated DR detection in Brazilian population, especially in screening campaigns with large-scale diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years with type 1 or 2 diabetes mellitus

Exclusion Criteria:

* Previous cataract, trabeculectomy or vitrectomy
* Aphakia
* External ocular infections
* Glaucoma (IOP of > 21 mmHg or regular use of more than 2 IOP lowering drugs)
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic retinopathy.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To compare the sensitivity and specificity of automated grading system versus human grading in detecting diabetic retinopathy | 6 months
  The aim of this study is to determine the sensitivity and specificity of automated grading system in detecting diabetic retinopathy compared with human grading on the population of annual massive screening campaign for diabetes conducted in the Northeast of Brazil.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Andrade, M.D., Study Director — Research Director
Locations (1):
- Retina Clinic, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mendes AB, Fittipaldi JA, Neves RC, Chacra AR, Moreira ED Jr. Prevalence and correlates of inadequate glycaemic control: results from a nationwide survey in 6,671 adults with diabetes in Brazil. Acta Diabetol. 2010 Jun;47(2):137-45. doi: 10.1007/s00592-009-0138-z. Epub 2009 Aug 5. PMID 19655083
- [Result] Soto-Pedre E, Navea A, Millan S, Hernaez-Ortega MC, Morales J, Desco MC, Perez P. Evaluation of automated image analysis software for the detection of diabetic retinopathy to reduce the ophthalmologists' workload. Acta Ophthalmol. 2015 Feb;93(1):e52-6. doi: 10.1111/aos.12481. Epub 2014 Jun 30. PMID 24975456
- [Result] Scotland GS, McNamee P, Philip S, Fleming AD, Goatman KA, Prescott GJ, Fonseca S, Sharp PF, Olson JA. Cost-effectiveness of implementing automated grading within the national screening programme for diabetic retinopathy in Scotland. Br J Ophthalmol. 2007 Nov;91(11):1518-23. doi: 10.1136/bjo.2007.120972. Epub 2007 Jun 21. PMID 17585001
- [Result] Fleming AD, Philip S, Goatman KA, Olson JA, Sharp PF. Automated assessment of diabetic retinal image quality based on clarity and field definition. Invest Ophthalmol Vis Sci. 2006 Mar;47(3):1120-5. doi: 10.1167/iovs.05-1155. PMID 16505050
- [Result] Malerbi FK, Morales PH, Farah ME, Drummond KR, Mattos TC, Pinheiro AA, Mallmann F, Perez RV, Leal FS, Gomes MB, Dib SA; Brazilian Type 1 Diabetes Study Group. Comparison between binocular indirect ophthalmoscopy and digital retinography for diabetic retinopathy screening: the multicenter Brazilian Type 1 Diabetes Study. Diabetol Metab Syndr. 2015 Dec 21;7:116. doi: 10.1186/s13098-015-0110-8. eCollection 2015. PMID 26697120
- [Result] Grading diabetic retinopathy from stereoscopic color fundus photographs--an extension of the modified Airlie House classification. ETDRS report number 10. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):786-806. PMID 2062513
- [Result] Ribeiro L, Oliveira CM, Neves C, Ramos JD, Ferreira H, Cunha-Vaz J. Screening for Diabetic Retinopathy in the Central Region of Portugal. Added Value of Automated 'Disease/No Disease' Grading. Ophthalmologica. 2014 Nov 26. doi: 10.1159/000368426. Online ahead of print. PMID 25427567
- [Result] Bhaskaranand M, Ramachandra C, Bhat S, Cuadros J, Nittala MG, Sadda S, Solanki K. Automated Diabetic Retinopathy Screening and Monitoring Using Retinal Fundus Image Analysis. J Diabetes Sci Technol. 2016 Feb 16;10(2):254-61. doi: 10.1177/1932296816628546. PMID 26888972